CLINICAL TRIAL: NCT03885232
Title: Presumptively Initiating Vaccines and Optimizing Talk With Motivational Interviewing (PIVOT With MI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Missouri, Kansas City (Other); Portland State University (Other); University of Washington (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH); Seattle Children's Hospital (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17-1274; 1R01HD093628-01A1 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-03-21 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Preventive Health Services (PREV HEALTH SERV)
Keywords: Communication; Immunization
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data Analysis study team members and parent participants will be masked to study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIVOT with MI (Experimental): Clinics in which the Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing (PIVOT-MI) communication strategy has been implemented.
  Interventions: Behavioral: Experimental: PIVOT with MI
- Control (Active Comparator): Clinics delivered standard care.
  Interventions: Other: Active Comparator: Control

INTERVENTIONS:
Behavioral: Experimental: PIVOT with MI — Providers in participating intervention clinics will be trained in the PIVOT-MI strategy in which a presumptive format is used to initiate the childhood vaccine recommendation with all parents followed by use of motivational interviewing (MI) with parents who voice resistance to that recommendation. Parent participants will receive PIVOT-MI.
  Arms: PIVOT with MI
Other: Active Comparator: Control — Providers at participating control clinics will deliver care as usual. Parent participants will receive standard care.
  Arms: Control

SUMMARY:
The overall goal of this project is to determine whether a novel and innovative provider communication strategy is effective in improving vaccine acceptance among vaccine-hesitant parents (VHPs) and visit experience among VHPs and their health care providers.

DETAILED DESCRIPTION:
The primary goal of this covariate constrained, cluster randomized controlled trial is to evaluate the effectiveness of an innovative provider communication strategy (PIVOT-MI) intervention in improving provider-parent vaccine discussions and increasing vaccine acceptance. Providers at intervention clinics will be trained to use the PIVOT-MI strategy in which a presumptive format is used to initiate the childhood vaccine recommendation with all parents, followed by use of motivational interviewing (MI) with parents who voice resistance to that recommendation. Providers at control clinics will deliver care as usual.

Specific aims are to evaluate the impact of PIVOT-MI, relative to control, on (1) child's immunization status; (2) parent-rated visit experience with their child's provider; and (3) change in provider experience of the vaccine discussion with vaccine-hesitant parents.

ELIGIBILITY:
Inclusion Criteria:

* Parents: must be English or Spanish speaking, ≥18 years old, have an infant ≤18 months old, have legal guardianship of the infant, and is receiving pediatric care at an enrolled clinic
* Providers: All providers at participating study practices will be eligible to participate.

Exclusion Criteria:

* Parents: not English or Spanish speaking, under 18 years old, have an infant older than 18 months, not the legal guardian of the infant, and/or having a child who is not receiving pediatric care at an enrolled clinic.
* Providers: Providers who are not at participating study practices.

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17446 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado, Denver; Douglas Opel, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Opel DJ, Robinson JD, Zhou C, Colborn K, Spielvogle H, Furniss A, Spina C, Perreira C, O'Leary ST. Tiered Clinician Vaccine Communication Strategy to Improve Childhood Vaccine Uptake: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e257814. doi: 10.1001/jamanetworkopen.2025.7814. PMID 40305020
- [Derived] Opel DJ, Robinson JD, Spielvogle H, Spina C, Garrett K, Dempsey AF, Perreira C, Dickinson M, Zhou C, Pahud B, Taylor JA, O'Leary ST. 'Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing' (PIVOT with MI) trial: a protocol for a cluster randomised controlled trial of a clinician vaccine communication intervention. BMJ Open. 2020 Aug 11;10(8):e039299. doi: 10.1136/bmjopen-2020-039299. PMID 32784263

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinics
Groups:
- PIVOT With MI: Clinics in which the Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing (PIVOT-MI) communication strategy was implemented.
Period: Overall Study
Arm/Group | PIVOT With MI | Control
Started | 9905; 12 clinics | 7541; 12 clinics
Participants Are Clinicians | 127; 12 clinics | 85; 12 clinics
Participants Are Parents Within the Parent/Infant Dyads | 4889; 12 clinics | 3728; 12 clinics
Participants Are Infants Within the Parent/Infant Dyads | 4889; 12 clinics | 3728; 12 clinics
Completed | 9799; 12 clinics | 7486; 12 clinics
Not Completed | 106; 0 clinics | 55; 0 clinics
Not completed — Lost to Follow-up | 74 | 32
Not completed — Staff turnover at enrolled clinics | 32 | 23

BASELINE CHARACTERISTICS:
Groups:
- Control: Care delivered as usual.
- Total: Total of all reporting groups
Arm/Group | PIVOT With MI | Control | Total
Number analyzed (Participants) | 9905 | 7541 | 17446
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was collected for parent/infant dyads, where all baseline characteristics refers to parents. Characteristics were not collected for infants. Age was not a measure collected for clinicians.
  Participants
    Parent/Infant Dyads: number analyzed (Participants) | 4889 | 3728 | 8617
    Parent/Infant Dyads: <=18 years | 0 | 0 | 0
    Parent/Infant Dyads: Between 18 and 65 years | 4889 | 3728 | 8617
    Parent/Infant Dyads: >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data was collected for parent/infant dyads, where all baseline characteristics refers to parents. Characteristics were not collected for infants. Population: Participants are split into two groups: parent/infant dyads and clinicians. Demographics for each group were collected separately, as their data is analyzed separately.
  Participants
    Parent/Infant Dyads: number analyzed (Participants) | 4889 | 3728 | 8617
    Parent/Infant Dyads: Female | 4138 | 3200 | 7338
    Parent/Infant Dyads: Male | 567 | 425 | 992
    Parent/Infant Dyads: Unknown | 184 | 103 | 287
    Clinicians: number analyzed (Participants) | 127 | 85 | 212
    Clinicians: Female | 88 | 61 | 149
    Clinicians: Male | 39 | 24 | 63
    Clinicians: Unknown | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data was collected for parent/infant dyads, where all baseline characteristics refers to parents. Characteristics were not collected for infants. Population: Participants are split into two groups: parent/infant dyads and clinicians. Demographics for each group were collected separately, as their data is analyzed separately.
  Participants
    Parent/Infant Dyads: number analyzed (Participants) | 4889 | 3728 | 8617
    Parent/Infant Dyads: Hispanic or Latino | 551 | 460 | 1011
    Parent/Infant Dyads: Not Hispanic or Latino | 4,162 | 3158 | 7320
    Parent/Infant Dyads: Unknown or Not Reported | 176 | 110 | 286
    Clinicians: number analyzed (Participants) | 127 | 85 | 212
    Clinicians: Hispanic or Latino | 3 | 5 | 8
    Clinicians: Not Hispanic or Latino | 123 | 79 | 202
    Clinicians: Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data was collected for parent/infant dyads, where all baseline characteristics refers to parents. Characteristics were not collected for infants. Population: Participants are split into two groups: parent/infant dyads and clinicians. Demographics for each group were collected separately, as their data is analyzed separately.
  Participants
    Parent/Infant Dyads: number analyzed (Participants) | 4889 | 3728 | 8617
    Parent/Infant Dyads: American Indian or Alaska Native | 62 | 28 | 90
    Parent/Infant Dyads: Asian | 228 | 358 | 586
    Parent/Infant Dyads: Native Hawaiian or Other Pacific Islander | 14 | 19 | 33
    Parent/Infant Dyads: Black or African American | 85 | 63 | 148
    Parent/Infant Dyads: White | 3997 | 2931 | 6928
    Parent/Infant Dyads: More than one race | 188 | 142 | 330
    Parent/Infant Dyads: Unknown or Not Reported | 315 | 187 | 502
    Clinicians: number analyzed (Participants) | 127 | 85 | 212
    Clinicians: American Indian or Alaska Native | 0 | 0 | 0
    Clinicians: Asian | 13 | 8 | 21
    Clinicians: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Clinicians: Black or African American | 0 | 1 | 1
    Clinicians: White | 106 | 74 | 180
    Clinicians: More than one race | 6 | 2 | 8
    Clinicians: Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants] — Participant totals include both parents, infants, and clinicians.
  participants
    United States | 9905 | 7541 | 17446

OUTCOME MEASURES:

1. Primary Outcome: Child Immunization Status at 19 Months, 0 Days of Age Characterized as Percent Days Under-immunized (DUI)
Description: Immunization status was obtained from WA or CO state immunization registry or directly from participating practices. At enrollment, parent/infant dyads completed the Parental Attitudes about Childhood Vaccines short version (PACV-SF), a validated survey scored from 0 to 4. A score of 2 or more represented parent/infant dyad with negative vaccine attitudes. Among parent/infant dyads with negative vaccine attitudes, the child's immunization status at 19 months was calculated based on recommended ages and intervals between doses provided by ACIP for summing late days for each dose of the 8 routine vaccines recommended by 19 months (HepB, rotavirus, DTaP, Hib, pneumococcal conjugate, inactivated polio virus, MMR, and varicella). There was a max of 23 recommended doses for the 8 vaccines - doses varied depending on brand. Total max DUI was a sum of total possible days late for each dose through 19mo(2830 days).Percent DUI was calculated by dividing child's DUI by the total maximum DUI.
Time Frame: Child's immunization status at 19 months of age
Population: Infants of parents/caregivers who had negative vaccine attitudes (Parental Attitudes about Childhood Vaccines short form (PACV-SF) score of 2 or higher)
Measure: Mean (Standard Deviation); unit: percentage of days under-immunized
Groups:
- PIVOT With MI: Parent/Caregiver and Infant Dyad: Parent/Caregiver and Infant dyads at participating clinics trained to use the Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing (PIVOT-MI) communication strategy.
- Control: Parent/Caregiver and Infant Dyad: Parent/Caregiver and Infant dyads at participating clinics in the control arm who received care as usual.
Arm/Group | PIVOT With MI: Parent/Caregiver and Infant Dyad | Control: Parent/Caregiver and Infant Dyad
Number analyzed (Participants) | 586 | 351
percentage of days under-immunized | 32 (38) | 24 (32)
Statistical Analysis 1: Comparison: PIVOT With MI: Parent/Caregiver and Infant Dyad vs Control: Parent/Caregiver and Infant Dyad; Test type: Superiority — We applied a mixed zero-inflated beta regression model that included a fixed binary factor for treatment arm, a random effect for clinic to account for correlation within clinics, and unbalanced parent demographics across study arms; p = 0.9, Generalized linear mixed effects regress; Generalized linear mixed effects regression models; Incidence Rate Ratio (IRR) = 1.04, 95% CI 2-sided [0.68 to 1.60]

2. Secondary Outcome: Post-Visit Parental Satisfaction Survey Scored on a 7-point Likert Scale
Description: To assess parental satisfaction with their clinician during a health supervision visit, we asked all vaccine hesitant parents (identified by a Parental Attitudes about Childhood Vaccines-Short Form (PAC-V SF) score of 2 or more) in both both intervention and control arms if they would complete an additional 15-question survey over the phone within 24-48 hours after the completion of a health supervision visit for their child around 6 months of age. Due to COVID-19 restrictions, we had to extend the time frame to within 1 week after a health supervision visit at 2, 4, or 6 months of age. Ratings were on a 7-point Likert scale - Very Poor (1), Poor (2), Fair (3), Good (4), Very Good (5), Excellent (6), Outstanding (7). Overall experience with a rating of "Good (4)" or higher was considered to be a satisfactory visit.
Time Frame: approximately 6 months post birth
Population: A subset of parent/infant dyads in both intervention and control clinics who were identified as vaccine hesitant (score of 2 or more on the Parental Attitudes about Childhood Vaccines short form (PACV-SF)) and who completed the post-healthcare visit satisfaction survey.
Measure: Number; unit: % of participants scoring 4 or higher
Arm/Group | PIVOT With MI: Parent/Caregiver and Infant Dyad | Control: Parent/Caregiver and Infant Dyad
Number analyzed (Participants) | 73 | 46
% of participants scoring 4 or higher | 96 | 96
Statistical Analysis 1: Comparison: PIVOT With MI: Parent/Caregiver and Infant Dyad vs Control: Parent/Caregiver and Infant Dyad; Calculated individual survey means for vaccine hesitant parents who participated in the survey. Survey consisted of 15 questions with a 7-point Likert scale. We then created a dichotomous variable where 1 = mean > or equal to 6; 0 = mean < 6; Test type: Superiority; p < 0.05, Chi-squared; Other = 1.0

3. Secondary Outcome: Change in Clinician Self-Efficacy With Parent/Infant Dyads With Negative Vaccine Attitudes - Pre-vs Post-Surveys
Description: To assess changes in clinicians' perceived self-efficacy when discussing vaccines with parents/infant dyads with negative vaccine attitudes, a survey was administered to all participating clinicians at baseline and at study completion asking about vaccine recommendation behaviors and how they perceived their impact on parental decision making regarding vaccines. Self-efficacy was assessed with a 3-part question scored on a Likert Scale - Strongly Disagree, Somewhat Disagree, Somewhat Agree, Strongly Agree. Changes in perceived self-efficacy over time was assessed by comparing the number of clinicians who answered "Strongly Agree" or "Somewhat Agree" to the statement "When parents wish to delay or refuse childhood vaccines for their child, there is not much I can say to change their minds" at baseline and at post-study. Note that fewer clinicians completed the post-study survey due to such factors as retirement and staff turnover.
Time Frame: At Baseline and Post-Intervention (up to 2 years after baseline)
Population: Clinicians enrolled across n=24 clinics (n=12 intervention clinics; n=12 control clinics)
Measure: Count of Participants; unit: Participants
Groups:
- PIVOT With MI: Clinicians: Clinicians at participating clinics randomized to the intervention arm and trained in the Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing (PIVOT-MI) communication strategy.
- Control: Clinicians: Clinicians at participating control clinics who delivered care as usual.
Arm/Group | PIVOT With MI: Clinicians | Control: Clinicians
Number analyzed (Participants) | 127 | 85
Participants
  Baseline Survey Results | 54 | 39
  Post-Study Survey Results: number analyzed (Participants) | 75 | 52
  Post-Study Survey Results | 23 | 20
Statistical Analysis 1: Comparison: PIVOT With MI: Clinicians vs Control: Clinicians; 1. Ho: No difference in the proportion of clinicians using presumptive and Motivational Interviewing techniques between intervention and control. 2. Ho: No difference in the proportion of clinicians time spent talking to vaccine hesitant parents between intervention and control; Test type: Superiority; p < 0.05, Generalized linear mixed effects regress; Adjusted for: study arm, study period (pre vs. post), years in practice, provider type, interaction between study arm and study period; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.66 to 5.64]

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: No adverse events collected
Groups:
- Control: Clinics delivered care as usual.
Arm/Group | PIVOT With MI | Control
All-Cause Mortality (participants affected / at risk) | 0/5016 | 0/3813
Serious Adverse Events (participants affected / at risk) | 0/5016 | 0/3813
Other Adverse Events (participants affected / at risk) | 0/5016 | 0/3813

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT03885232/Prot_SAP_000.pdf